CLINICAL TRIAL: NCT05845528
Title: Impact of Susceptibility to Placebo on the Effect of Transcranial Direct Current Stimulation (tDCS) in Fibromyalgia: a Randomized Clinical Trial With Extended Home Stimulation
Brief Title: Impact of Susceptibility to Placebo on the Effect of Transcranial Direct Current Stimulation (tDCS) in Fibromyalgia
Acronym: FIBROTEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200383
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; tDCS; placebo effect; pain; b-endorphin
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Parallel Group, Sham-Controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The researcher will receive equipment already programmed by a research assistant, so the researcher who will deliver the tDCS to perform stimulation will not know the programed stimulation. Patients will be instructed to discuss aspects of treatment with the respective investigator. Two independent evaluators who will not participate in the consultations where guidance on the use of tDCS will be provided will be trained to make outcome assessments in follow-up. Patients will not be aware of the type of intervention received, since the sham condition produces a stimulus, but no expected effects. In order to study the level of the blinding, at each moment of evaluation, the patient will be asked about the type of intervention that he / she believes to have received (active or simulated), and about the degree of safety in the response, using a standardized questionnaire. The blinding will be evaluated at the end of each treatment week by means of a standardized instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respondres placebo effect (Placebo Comparator): Intervention: 'Transcranial Direct Current Stimulation - tDCS
  * The patients will receive tDCS stimulation treatment prefrontal cortex dorso lateral
  * According to 10-20 EEG system, anode will be placed at left F3 and cathode at contralateral F4.
  * Placebo stimulation uses a 2 milliamperes current during in the first minutes, in the 10 min and in 19 minutes.
  Interventions: Device: s-tDCS; Device: a- tDCS
- No respondres placebo effect (Active Comparator): Intervention: 'Transcranial Direct Current Stimulation - tDCS
  * The patients will receive tDCS stimulation treatment prefrontal cortex dorso lateral
  * According to 10-20 EEG system, anode will be placed at left F3 and cathode at contralateral F4.
  * Active stimulation uses a 2 milliamperes current during 20 minutes.
  Interventions: Device: s-tDCS; Device: a- tDCS

INTERVENTIONS:
Device: s-tDCS — - Intervention: tDCS is a therapeutic method that modulates the membrane potential, where anodic stimuli induce cortical excitability and cathodic stimuli reduce it
Device: a- tDCS — - Intervention: tDCS is a therapeutic method that modulates the membrane potential, where anodic stimuli induce cortical excitability and cathodic stimuli reduce it

SUMMARY:
Fibromyalgia (FM) is a syndrome characterized by generalized musculoskeletal pain, fatigue, non-restorative sleep, cognitive changes, depressive and neurovegetative symptoms. It is known that conventional pharmacological therapies produce responses with little clinical impact in more than 50% of patients. Functional alterations of the motor cortex and its connections with subcortical structures have also been demonstrated in FM. Based on the above, the objective of this research is to identify subgroups of patients with greater potential for responsiveness to treatment with a view to advancing diagnosis and treatment. In this study, the therapeutic target will be transcranial direct current stimulation (tDCS) according to the potential of responsiveness to the placebo effect, with the precise location of the stimulation area by a neuronavigation system, with the objective of counter-regulating the dysfunctional processes responsible for triggering and maintaining FM symptoms. Therefore, this clinical trial aims to compare the efficacy of anodal tDCS applied to the left dorsolateral prefrontal cortex (DLPFC) compared to simulated tDCS in FM, according to susceptibility to placebo effect and serum endorphin levels.

DETAILED DESCRIPTION:
This is clinical trial aims to compare the efficacy of anodal tDCS applied to the left dorsolateral prefrontal cortex (DLPFC) compared to simulated tDCS in FM, according to susceptibility to placebo effect and serum endorphin levels, in the following outcomes (1) treatment effectiveness, which includes daily measures recorded in an application by the Brief Pain Inventory (BPI), which allows pain assessment from a multidimensional perspective (pain intensity and interference in general activities, mood, mobility, work, personal relationships, sleep and enjoyment of life, etc.) (primary outcome). Secondary outcomes: the impact of pain on quality of life; levels of depressive symptoms; (2) Outcomes in psychophysical measures: pain threshold to electrical stimulation and heat; temporal summation to electrical stimulus; descending pain modulatory system function; (3) Identify predictors of response to the placebo effect through a hierarchical model with an analytical structure defined a 'priori', considering the hierarchical relationships between potential predictors such as: disability due to pain, catastrophism, depressive symptoms, psychiatric diagnoses, level of central sensitization, endorphin serum levels at baseline, drugs in use, etc. In this randomized, controlled, sham-controlled, parallel, double-blind clinical trial, 84 women with FM will be included, according to the criteria of the American College of Rheumatology (2016), aged between 18 and 70 years. Patients will be submitted to a simulated tDCS face-to-face session, mounted on the left DLPFC, and with a variation presented in the Numerical Verbal Pain Scale (NPS 0-10) equal to or greater than thirty percent of the baseline, the patient will be considered a high responder and below this low responder rate. This will be the criterion used to stratify randomization. They will receive 30 sessions of anodal tDCS lasting 20 min, with a current of 2 mA, applied to the left DLPFC at home. The location of the stimulation area will be done by a neuronavigation system. Patients will receive training in using the tDCS equipment.

They will have access to an instructional video on tDCS and a way of communicating with the team through Whatsapp. The follow-up time after the end of stimulation will be 12 weeks as recommended by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT). Patients should respond daily to BPI and possible side effects of tDCS. Home tDCS will be carried out with equipment developed by our research group, in partnership with Biomedical Engineering at Hospital de Clínicas de Porto Alegre (HCPA), with patent registration with the National Institute of Industrial Property (INPI) under number BR2020150164500. Our hypothesis is that active tDCS has a greater effect than simulated tDCS and that stimulation on the DLPFC has a greater impact in patients with greater responsiveness to the placebo effect on psychological symptoms, functional capacity for activities of daily living and inhibitory modulatory system function. descendant of pain. It is expected that the level of cortical disinhibition assessed by TMS measurements, as well as serum ß-endorphin levels, can serve as predictors of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 65 years; who can read and write, with a confirmed diagnosis of FM according to the American College of Rheumatology criteria (2010-2016). Pain score equal to or greater than six on the Numerical Pain Scale (NPS 0-10) on most days of the last 3 months.

Exclusion Criteria:

* Residing outside the greater Porto Alegre area and pregnancy. Contraindications to TMS and tDCS: metallic implant in the brain; medical devices implanted in the brain, cardiac pacemakers; cochlear implant; history of alcohol or drug abuse in the last 6 months; neurological pathologies; hx of head trauma or neurosurgery; decompensated systemic diseases and chronic inflammatory diseases (lupus, rheumatoid arthritis, Reiter's syndrome); uncompensated hypothyroidism; personal history of cancer, past or undergoing treatment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
1.Change in pain level - first phase | Time Frame: 1 month
  Change from before and after the First phase of treatment on Pain scores assessed by a Numerical Pain Scale (NPS 0 to 10) (0 means no pain - 10 means the worst pain imaginable)
Change in functional capacity - first phase | 1 month
  The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning

SECONDARY OUTCOMES:
Change in pain level - second phase | 3 months
  Change from before and after the Second phase of treatment on Pain scores assessed by a visual analogue scale (VAS 0 to 100mm) (0 means no pain - 100 means the worst pain imaginable)
Change in functional capacity - second phase | 3 months
  Change from before and after the First phase of treatment on Total score on the Brazilian Profile of Chronic Pain: Screen (BPCP:S) (range from 0 to 93; high numbers means more pain severity, interference in daily activities and emotional burden)
Change in Function of modulatory descending system | 1 month
  Change from before and after the First phase of treatment on the score in a numerical pain scale (NPS 0-10) for a moderate heat pain stimulus to the right arm (ventral region) during a conditioned pain modulation task (CPM-task), where participant keeps the counter-lateral hand in an iced cold water (0 to 1º Celsius)
Change in Function of corticospinal pathway | Time Frame: 1 month
  Change from before and after the First phase of treatment on measures of motor threshold (MT), motor evoked potential (MEP), intracortical facilitation (ICF), short intracortical inhibition (SICI), and cortical silent period (CSP) assessed with transcranial magnetic stimulation (TMS).
7. Change in levels of Brain derived neurotrophic factor - BDNF | Time Frame: 1 month
  Blood samples will be collected at baseline and after the First phase of intervention in order to determine BDNF serum levels using a standardized kit

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clauw DJ, Arnold LM, McCarberg BH; FibroCollaborative. The science of fibromyalgia. Mayo Clin Proc. 2011 Sep;86(9):907-11. doi: 10.4065/mcp.2011.0206. PMID 21878603
- [Background] Keeser D, Meindl T, Bor J, Palm U, Pogarell O, Mulert C, Brunelin J, Moller HJ, Reiser M, Padberg F. Prefrontal transcranial direct current stimulation changes connectivity of resting-state networks during fMRI. J Neurosci. 2011 Oct 26;31(43):15284-93. doi: 10.1523/JNEUROSCI.0542-11.2011. PMID 22031874
- [Background] Zanette SA, Dussan-Sarria JA, Souza A, Deitos A, Torres IL, Caumo W. Higher serum S100B and BDNF levels are correlated with a lower pressure-pain threshold in fibromyalgia. Mol Pain. 2014 Jul 8;10:46. doi: 10.1186/1744-8069-10-46. PMID 25005881
- [Derived] Caumo W, Franca BR, Orzechowski R, Bueno G, Franca de Souza A, Dos Santos da Silva JV, Sanches PRS, Da Silva DP Jr, Torres ILS, Hirakata VN, Pacheco-Barrios K, Fregni F. Home-Based Transcranial Direct Current Stimulation vs Placebo for Fibromyalgia: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2514262. doi: 10.1001/jamanetworkopen.2025.14262. PMID 40478572